CLINICAL TRIAL: NCT01669421
Title: Effect of a Higher Dose of Alpha-1 Antitrypsin Augmentation Therapy on Lung Inflammation in Subjects With Alpha-1 Antitrypsin Deficiency.
Brief Title: Effect of Double Dose of Alpha 1-antitrypsin Augmentation Therapy on Lung Inflammation.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Campos, MD (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor-Investigator, Michael Campos, MD, Associate Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20100844
Record Dates: First submitted 2012-08-14; First posted 2012-08-21 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Alpha 1 Antitrypsin Deficiency
Keywords: Alpha 1
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alpha-1 Antitrypsin (human) standard dose baseline (Experimental): Alpha-1 Antitrypsin (human) 60 mg per kg per week for 4 weeks. Study week 4
  Interventions: Drug: Alpha-1 Antitrypsin (human)
- Alpha-1 Antitrypsin (human) Double dose (Experimental): Alpha-1 Antitrypsin (human) 120 mg/kg per week for 4 weeks. Study week 8
  Interventions: Drug: Alpha-1 Antitrypsin (human)
- Alpha-1 Antitrypsin (human) standard dose (Experimental): 4 weeks on A1PI at 60 mg/kg per week after the other 2 phases. Collected@ study week 12
  Interventions: Drug: Alpha-1 Antitrypsin (human)

INTERVENTIONS:
Drug: Alpha-1 Antitrypsin (human) — Comparison of Zemaira (Alpha 1 Antitrypsin Human) 120 mg/kg/weekly for four weeks versus 2 phases with same drug administered at standard doses of 60 mg/kg/weekly for four weeks each
  Other Names: Zemaira; Alpha-1 proteinase inhibitor (human)

SUMMARY:
The current treatment of individuals with alpha-1 antitrypsin deficiency (AATD) who develop lung disease (COPD) is the administration of intravenous purified alpha-1 antitrypsin (augmentation therapy) at a fixed dose of 60 mg/kg per week. This dose aims at increasing the deficient AAT serum levels just above a predetermined "safety threshold" of 11 uM. However, normal levels of AAT are between 25-50 uM.

AAT has shown not only to inhibit lung proteases such as neutrophil elastase, but also to modulate inflammation. Given that many subjects with AATD who receive augmentation therapy still have significant lung disease and inflammation, this study will evaluate whether doubling the dose to 120 mg/kg/week has an effect in decreasing lung inflammation.

Only the dosing of 60 mg/kg /week has received FDA approval. FDA has granted an IND number to this study to test the higher dose of 120 mg/kg/week.

The study will evaluate systemic (serum) and pulmonary (bronchoscopy samples)markers of inflammation in 3 phases: standard dose (4 weeks), double dose (4 weeks) and standard dose (4 weeks).

DETAILED DESCRIPTION:
This is a pilot study to test the effect of double dose augmentation therapy with Zemaira (CSL Behring) on lung inflammation, compared with standard doses of 60 mg/kg/week.

Our hypothesis is that some patients with AATD receiving augmentation therapy at the standard dose of 60 mg/kg/week continue to have a significant lung inflammation that may lead to detrimental clinical consequences. This inflammation can be further reduced with higher AAT dosing.

The study will enroll 20 subjects with AATD and COPD already receiving augmentation therapy with any brand at standard doses for at least a month. For inclusion and exclusion criteria see below.

Protocol:

The study will take place over approximately 12 weeks: a month receiving Zemaira at standard dose (60 mg/kg/week), a month at double dose (120 mg/kg/week) and a month at standard dose (60 mg/kg/week). The infusions at standard doses will be done at home and infusions with higher doses will be provided at the study site.

the study involves scheduled blood draws for clinical labs and serum for research samples. At the end of each phase a bronchoscopy will be performed (3 in total) to obtain research samples (lung lavage, brushings and endobronchial biopsies).

The first bronchoscopy after receiving 4 weeks of standard augmentation therapy will assess the "residual" inflammation that may be present despite augmentation therapy. The second bronchoscopy after double dose augmentation therapy phase will be to assess changes (decreases) in inflammatory markers. The third bronchoscopy after resuming standard dosing is to assess if inflammation returned to baseline levels (required for proof of concept).

There will be approximately 9 visits to the study clinic. This study does not include placebo (no active drug) treatment. Besides blood draws and bronchoscopy, the study will include questionnaires and lung function testing.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females aged between 18 and 75 years.
* Diagnosis of AATD, based on documentation of "at-risk" genotypes such as Pi ZZ, SZ or Znull OR documentation of a pre-therapy AAT level < 11 µM.
* Evidence of COPD (emphysema or airflow obstruction) with FEV1 < 80%
* Receiving standard dose of augmentation therapy (with any commercial formulation) for at least 1 month at the dose of 60 mg/kg/week.
* At least ONE of the following criteria of disease severity:

  * 2 or more acute exacerbations or 1 hospitalization due to respiratory symptoms in the past 12 months. Definition of exacerbations: the use of antibiotics and a course of steroids to treat a flare of pulmonary symptoms, regardless if the subject required emergency room care or hospital admission. The diagnosis of the acute exacerbation will be obtained by direct history obtained from the patient and confirmed by the PI. Attempts should be made to have documentation from the patient's treating physicians, although not required for study entry.
  * St. George Respiratory Questionnaire (SGRQ) total score ≥ 60.
  * Chronic bronchitis: daily or almost daily sputum expectoration at least 3 months of the year for at least 2 consecutive years. The diagnosis of chronic bronchitis will be obtained by direct history obtained from the patient and confirmed by the PI. Attempts should be made to have documentation from the patient's treating physicians, although not required for study entry.
  * Documented FEV1 decline of at least ≥ 60 ml/year for 2 consecutive years while receiving augmentation therapy

Exclusion Criteria:

- Patients unsuitable to have a bronchoscopy due to poor clinical condition as judged by the PI. In general we will exclude subjects with hypoxemia, coagulopathy or FEV1 below 40% predicted.

Note: Subjects with FEV1 values below 40% predicted may be included and reassessed after optimization of therapy. Final determination to include the patient if deemed suitable for the procedure will be determined by the PI before first planned bronchoscopy (regardless of FEV1 value).

* Patients participating in other clinical trials.
* Use of chronic antibiotics or oral steroids
* Continues to smoke
* Inability to sign informed consent
* Pregnancy or willing to become pregnant
* Known IgA deficiency (we will include only patients already receiving augmentation therapy so it will be unlikely to encounter this exclusion criteria)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Campos, MD, Principal Investigator — University of Miami
Locations (1):
- Division of Pulmonary and Critical Care, Human Reseach, U of Miami, Miami, Florida, United States

REFERENCES:
- [Background] Tonelli AR, Brantly ML. Augmentation therapy in alpha-1 antitrypsin deficiency: advances and controversies. Ther Adv Respir Dis. 2010 Oct;4(5):289-312. doi: 10.1177/1753465810373911. Epub 2010 Jul 22. PMID 20650978
- [Background] Stockley RA, Bayley DL, Unsal I, Dowson LJ. The effect of augmentation therapy on bronchial inflammation in alpha1-antitrypsin deficiency. Am J Respir Crit Care Med. 2002 Jun 1;165(11):1494-8. doi: 10.1164/rccm.2109013. PMID 12045122
- [Background] Petrache I, Hajjar J, Campos M. Safety and efficacy of alpha-1-antitrypsin augmentation therapy in the treatment of patients with alpha-1-antitrypsin deficiency. Biologics. 2009;3:193-204. doi: 10.2147/btt.2009.3088. Epub 2009 Jul 13. PMID 19707408
- [Derived] Campos MA, Geraghty P, Holt G, Mendes E, Newby PR, Ma S, Luna-Diaz LV, Turino GM, Stockley RA. The Biological Effects of Double-Dose Alpha-1 Antitrypsin Augmentation Therapy. A Pilot Clinical Trial. Am J Respir Crit Care Med. 2019 Aug 1;200(3):318-326. doi: 10.1164/rccm.201901-0010OC. PMID 30965011

RESULTS

PARTICIPANT FLOW:
Groups:
- Studied Population: All patients belong to one study arm. First they received standard dose augmentation therapy (60 mg/kg/week) x 4 weeks, then they receive experimental double dose (120 mg/kg/week) x 4 weeks and finally return to standard dose (60 mg/kg/week) for 4 additional weeks.
Period: Phase 1: Standard Dose Therapy
Arm/Group | Studied Population
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Period: Phase 2: Double Dose Therapy
Arm/Group | Studied Population
Started | 8
Completed | 8
Not Completed | 0
Period: Phase 3: Standard Dose Therapy
Arm/Group | Studied Population
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Alpha-1 Antitrypsin (Human): Alpha-1 Antitrypsin (human) 120 mg per kg per week for 4 weeks
  Alpha-1 Antitrypsin (human): Comparison of Zemaira (Alpha 1 Antitrypsin Human) 120 mg/kg/weekly for four weeks versus 2 phases with same drug administered at standard doses of 60 mg/kg/weekly for four weeks each
Arm/Group | Alpha-1 Antitrypsin (Human)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Changes in Inflammatory Biomarkers in Bronchoalveolar Lavage Fluid
Description: Assess the variations in the levels of several cytokines and inflammatory biomarkers in BAL after changing A1PI dosing.
  Measures were done using the bead technology.
Time Frame: Between baseline (week 4), double dose A1PI (week 8) and again standard dose (week 12)
Population: Subjects with AATD and COPD that require augmentation therapy
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Alpha-1 Antitrypsin (Human) Standard Dose Baseline | Alpha-1 Antitrypsin (Human) Double Dose | Alpha-1 Antitrypsin (Human) Standard Dose
Number analyzed (Participants) | 8 | 8 | 8
pg/ml
  IL-2 | 14.3 (7.3) | 8.1 (3.1) | 10.3 (1.7)
  IL-8 | 379.9 (294.3) | 563.2 (317.8) | 412.2 (160.1)
  IL-17 | 79.0 (27.8) | 61.5 (15.8) | 67.4 (8.5)
  BASIC FGF | 20.7 (9.3) | 15.4 (4.3) | 16.5 (2.1)
  GM-CSF | 114.9 (36.2) | 89.1 (33.6) | 105.4 (20.8)
  IL-15 | 116.5 (68.4) | 92.5 (38.9) | 90.5 (16.6)
  IL1alpha | 30.7 (18.7) | 27.4 (18.8) | 27.7 (6.0)
  IL-18 | 9.1 (7.4) | 8.1 (2.0) | 7.7 (1.6)
  M-CSF | 43.1 (18.9) | 37.0 (33.4) | 33.1 (19.4)
  IL-4 | 3.1 (0.6) | 3.0 (0.5) | 2.9 (0.4)
  IL-9 | 24.9 (4.8) | 23.1 (4.1) | 23.5 (3.3)
  Eotaxin | 154.0 (37.7) | 150.9 (44.6) | 138.0 (16.3)
Statistical Analysis 1: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose; IL-2; Test type: Other — Data was analyzed with multiple repeat ANOVA for all visits and paired samples were also evaluated; p < 0.05, Kruskal-Wallis
Statistical Analysis 2: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; IL-4; Test type: Other — Kruskal-Wallis; p = 0.035, Kruskal-Wallis
Statistical Analysis 3: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; IL-8; Test type: Other; p = 0.33, Kruskal-Wallis
Statistical Analysis 4: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; IL-9; Test type: Other; p = 0.68, Kruskal-Wallis
Statistical Analysis 5: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; IL-17; Test type: Other; p = 0.020, Kruskal-Wallis
Statistical Analysis 6: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; FGF; Test type: Other; p = 0.021, Kruskal-Wallis
Statistical Analysis 7: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; Eotaxin; Test type: Other; p = 0.02, Kruskal-Wallis
Statistical Analysis 8: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; GM-CSF; Test type: Other; p = 0.045, Kruskal-Wallis
Statistical Analysis 9: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; IL15; Test type: Other; p = 0.47, Kruskal-Wallis
Statistical Analysis 10: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; IL-1a; Test type: Other; p = 0.90, Kruskal-Wallis
Statistical Analysis 11: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; IL18; Test type: Other; p = 0.80, Kruskal-Wallis
Statistical Analysis 12: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; M-CSF; Test type: Other; p = 0.027, Kruskal-Wallis

2. Secondary Outcome: Change in Inflammatory Biomarkers in Serum Samples
Description: Assess the variations in the levels of cytokines and inflammatory biomarkers using the bead technology.
Time Frame: Between baseline (week 4), double dose A1PI (week 8) and again standard dose (week 12)
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Alpha-1 Antitrypsin (Human) Standard Dose Baseline: Alpha-1 Antitrypsin (human) 60 mg per kg per week for 4 weeks
- Alpha-1 Antitrypsin (Human) Double Dose: A1PI at 120 mg/kg per week for 4 weeks after subjects received 4 weeks standard dose
Arm/Group | Alpha-1 Antitrypsin (Human) Standard Dose Baseline | Alpha-1 Antitrypsin (Human) Double Dose | Alpha-1 Antitrypsin (Human) Standard Dose
Number analyzed (Participants) | 8 | 8 | 8
pg/ml
  IL-2 | 127.3 (114.0) | 114.5 (81.6) | 66.11 (95.7)
  IL-6 | 232.3 (212.0) | 222.4 (202.2) | 132.56 (161.0)
  IL-1beta | 11.2 (11.6) | 9.1 (7.7) | 34.06 (73.3)
  IL-4 | 14.5 (11.6) | 13.3 (9.4) | 9.73 (11.6)
  IL-10 | 85.8 (86.3) | 72.9 (58.1) | 50.62 (74.5)
  IFNy | 67.4 (67.9) | 67 (49.1) | 48.9 (63.6)
  CRP | 476.7 (358.9) | 1082.9 (1971.9) | 494.5 (453.1)
Statistical Analysis 1: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; No power calculation and this is an exploratory pilot analysis We expected cytokines to decrease after subjects receive double dose and a rebound after administering standard dose; Test type: Other; p = 0.07, Kruskal-Wallis

3. Secondary Outcome: Number of Adverse Events Reported
Time Frame: From Week 1 to week 12
Measure: Number; unit: Events
Groups:
- Alpha-1 Antitrypsin (Human) Standard Dose: 60 mg/kg per week after the prior 2 phases
Arm/Group | Alpha-1 Antitrypsin (Human) Standard Dose Baseline | Alpha-1 Antitrypsin (Human) Double Dose | Alpha-1 Antitrypsin (Human) Standard Dose
Number analyzed (Participants) | 10 | 8 | 8
Events | 0 | 0 | 0

4. Other Pre Specified Outcome: Elastin Degradation in BAL
Description: Desmosine/isodesmosine measured using mass spectometry.
Time Frame: Week 4 vs Week 8 vs Week 12
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Alpha-1 Antitrypsin (Human) Standard Dose Baseline: Alpha-1 Antitrypsin (human) 60 mg/kg per week for 4 weeks (measure at week 4)
- Alpha-1 Antitrypsin (Human) Double Dose: A1PI at 120 mg/kg per week x 4 weeks (measure at week 8)
- Alpha-1 Antitrypsin (Human) Standard Dose: A1PI at 60 mg/kg per week after double dose (measured at week 12)
Arm/Group | Alpha-1 Antitrypsin (Human) Standard Dose Baseline | Alpha-1 Antitrypsin (Human) Double Dose | Alpha-1 Antitrypsin (Human) Standard Dose
Number analyzed (Participants) | 8 | 8 | 8
ng/ml | 156.7 (103.2) | 62.89 (23.55) | 56.88 (25.46)
Statistical Analysis 1: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; Desmosine (DES) and isodesmosine (IDES) are used as indicator of elastin degradation. Levels of DES/IDES were measured using high-performance liquid chromatography and tandem mass spectrometry; Test type: Other — between Week 4 and Week 8; p = 0.03, t-test, 2 sided
Statistical Analysis 2: Comparison: Alpha-1 Antitrypsin (Human) Double Dose vs Alpha-1 Antitrypsin (Human) Standard Dose; between Week 8 and Week 12; Test type: Other; p = 0.33, t-test, 2 sided
Statistical Analysis 3: Comparison: Alpha-1 Antitrypsin (Human) Standard Dose Baseline vs Alpha-1 Antitrypsin (Human) Standard Dose; between Week 4 and Week 12; Test type: Other; p = 0.029, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Adverse event was recorded for each subject from study enrollment (day 0) through study end which was on the day of the last bronchoscopy at the end of phase 3 (week 12). Each subject was assessed weekly by phone calls and in-person at the end of each phase (day of bronchoscopies).
Groups:
- Phase 1: Standard Dose: Standard dose (60 mg/kg/week) Weeks1-4
- Phase 2: Double Dose: Double dose (120 mg/kg/week) weeks 4-8
- Phase 3: Standard Dose: Standard dose (60 mg/kg/week) weeks 8-12
Arm/Group | Phase 1: Standard Dose | Phase 2: Double Dose | Phase 3: Standard Dose
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/10 | 0/8 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Standard Dose (N=10) | Phase 2: Double Dose (N=8) | Phase 3: Standard Dose (N=8)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — 1 patient developed mild hemoptysis after bronchoscopy # 1 and withdrew from study
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — 1 patient developed respiratory distress after bronchoscopy # 1 and PI withdrew pt from study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No